CLINICAL TRIAL: NCT04577209
Title: Pediatric Source Control for Hazardous Particulate Exposure in Aerosol Generating Procedures
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants were enrolled due to unavailability of research staff.
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Chi-Ho Ban Tsui, Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 57866
Record Dates: First submitted 2020-09-28; First posted 2020-10-06 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Risk Reduction
Keywords: aerosol particles; anesthesia
MeSH Terms: conditions — Risk Reduction Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Pediatric Patients (Experimental): Participants undergoing anesthesia-related aerosol generating medical procedures (AGMPs) and pediatric otolaryngologic surgeries will have a local exhaust ventilation system to the exposure seen by the medical providers during the AGMPs and surgeries.
  Interventions: Device: Disposable oxygen face tent

INTERVENTIONS:
Device: Disposable oxygen face tent — Disposable oxygen face tent used to minimize aerosol particles (through suction) during aerosol generating anesthesia procedures.

SUMMARY:
There are two purposes of this study. The first purpose is to determine the exposure seen by medical providers (e.g. anesthesiologists, surgeons, and nurses) to infectious and smoke particulates generated during anesthesia-related aerosol generating medical procedures (AGMPs) and pediatric otolaryngologic surgeries (with and without an intubated airway). The second goal of this study is to apply a local exhaust ventilation system (LEVS) to re-evaluate the exposure seen by the same medical providers during the same AGMPs and surgeries.

DETAILED DESCRIPTION:
Prior to the patient entering the OR, particle counters (Digital PM2.5 Air Quality detector, ExGizmo, China) will ensure that the OR air quality has undergone the appropriate airflow exchanges and thus will all read 0.

Measurements will be taken every 30 seconds. A research assistant in the periphery of the OR will observe and record the following events: patient entrance into the OR, initiation of mask induction, intubation, rotation of OR table for surgery, initiation of surgery, completion of surgery, rotation of OR back to anesthesia, extubation, and patient departure from the OR. The particle counters will be positioned accordingly: 1) at the level of the patient's head, 2) at the level of the anesthesiologist/surgeon performing the AGMPs, 3) to the right of the patient, 4) to the left of the patient, 5) at the anesthesia workstation, and 6) at the circulating nurse's computer in the corner of the room. The particle counters will continue with measurements until the patient exits the OR. For patients randomized to the LEVS group, active suction will be provided through the use of a closed biohazardous smoke evacuation system (Neptune 3, Stryker, Michigan, USA) equipped with an internal high efficiency particulate air (HEPA) filter capable of capturing aerosolized particles as small as 0.1 mm with 99.99% efficiency via suction power up to 25 cubic feet per minute air exchange. The active suction will be positioned near the patient's airway without interfering with the AGMP, and across from the location of the anesthesiologist or surgeon performing the AGMP such that no HCW is positioned between the patient's airway and the suction device.

ELIGIBILITY:
Inclusion Criteria:

* children receiving anesthesia-related aerosol generating medical procedures

Exclusion Criteria:

* patients with positive COVID symptoms
* positive preoperative COVID testing

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Aerosolized particle concentration in air | Up to 60 minutes
  To measure the particle concentrations in the air (μg/m^3), particle counters will be located at each of the different healthcare worker positions in the operating room (OR) during an aerosol generating procedure either with a local evacuation system or without one. Measurements will be taken every 30 seconds from prior to the patient entering the OR to patient departure from the OR.

CONTACTS AND LOCATIONS:
Overall Officials: Ban C Tsui, MD, Study Director — Stanford University; Stephanie Pan, MD, Principal Investigator — Stanford University
Locations (1):
- Lucile Packard Childrens Hospital, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No